CLINICAL TRIAL: NCT04897126
Title: Efficacy and Safety of Shexiang Baoxin Pill in Patients With Ischemia With Non-Obstructive Coronary Artery: A Phase 4, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety of Shexiang Baoxin Pill in Patients With Ischemia With Non-Obstructive Coronary Artery
Acronym: LESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Collaborators: Shanghai Changzheng Hospital (Other); The Second People's Hospital Of Bengbu (Unknown); The Second Affiliated Hospital of Jiaxing University (Other); Zibo Municipal Hospital (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); Shanxi Cardiovascular Hospital (Other); The First Hospital of Hebei Medical University (Other); Tangshan Central Hospital (Other); Tie Fa Coal Group Ceneral Hospital of Liaoning Health Industry Group (Unknown); Ceneral Hospital Of Benxi Iron And Steel of Liaoning Health Industry Group (Unknown); General Hospital of Fuxin Mining Industry Group of Liaoning Health Industry Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LESS202010
Record Dates: First submitted 2021-05-19; First posted 2021-05-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Ischemia With Non-Obstructive Coronary Artery; Angina Pectoris; Coronary Heart Disease; X Syndrome, Angina
Keywords: Shexiang Baoxin Pill; MUSKARDIA; patients with chest pain due to non obstructive coronary artery disease
MeSH Terms: conditions — Angina Pectoris; Coronary Disease; Microvascular Angina

STUDY DESIGN:
Intervention Model Description: 1:1 stratified block random grouping according to the center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): The experimental group was treated with Shexiang Baoxin pill（MUSKARDIA） (4 pills / day, 3 times / day) on the basis of conventional treatment until the end of follow-up
  Interventions: Radiation: Shexiang Baoxin pill（MUSKARDIA）
- Placebo group (Placebo Comparator): The control group was given placebo（ 4 capsules / day, 3 times / day）on the basis of conventional treatment until the end of follow-up.
  Interventions: Radiation: Placebo

INTERVENTIONS:
Radiation: Shexiang Baoxin pill（MUSKARDIA） — On the basis of routine treatment, MUSK Pills were added to 4 capsules / day, 3 times per day until the end of follow-up.
  Other Names: routine treatment
  Arms: Experimental group
Radiation: Placebo — On the basis of routine treatment, Placebo were added to 4 capsules / day, 3 times per day until the end of follow-up.
  Other Names: routine treatment
  Arms: Placebo group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled clinical trial. Patients were treated with the trial drug or placebo in a 1:1 ratio. The control group was treated with placebo 4 pills / day, 3 times / day on the basis of conventional treatment until the end of follow-up, while the experimental group was treated with MUSK Pill 4 pills / day, 3 times / day on the basis of conventional treatment until the end of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The age was 18-75 years old, and the gender was not limited;
* The clinical diagnosis of angina pectoris or angina pectoris equivalent symptoms (attack at least twice a week), Within 1 year, coronary CTA or coronary angiography examination of coronary artery normal or lesions < 50%;
* Willing to follow up and sign informed consent.

Exclusion Criteria:

* Patients were selected and had no angina pectoris without medication
* History of vascular reconstruction within 6 months, CABG or PCI;
* Preparation for CABG or PCI during the trial period
* The maximum lesions of major branches of major vessels were ≥ 50% in CTA or angiographic examination;
* Severe cardiovascular and pulmonary vascular diseases: stubborn heart failure or cardiogenic shock, hypertrophic obstructive cardiomyopathy, severe aortic stenosis, incomplete closure, aortic dissection, pulmonary embolism;
* There were three months of acute myocardial infarction;
* Severe respiratory disease, COPD or active pulmonary infection;
* Although the patients with poor blood pressure control were treated with hypertension, the hypertension was not controlled and / or systolic pressure ≥ 180mmhg and diastolic pressure ≥ 110mmhg before the end of screening period;
* Severe liver and kidney diseases, such as liver and kidney dysfunction (alt, AST ≥ 1.5 times of the upper limit of normal value, Cr > 1.5 times of normal value), active liver disease, cirrhosis or uremia patients;
* Any other serious diseases or conditions such as malignant tumor, severe anemia, severe renal artery stenosis, severe anxiety depression (HAMD-17) and suicide or maniac mental illness;
* Participated in other clinical studies within 30 days before the selection, or is currently participating in other clinical studies;
* Pregnant, lactating women and women and men with recent birth plans;
* Allergic constitution or allergy to known components of the study drug;
* The researchers judged that the patients who were not suitable for the study were not suitable.

(Note: patients need to stop using other cardiovascular traditional Chinese patent medicines and simple preparations or traditional Chinese medicine for 7 days before enrollment.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Changes of Seattle angina pectoris scale | 12 weeks ± 1 week
  Main evaluation indicators

SECONDARY OUTCOMES:
Average number of angina attacks per week | 12 weeks ± 1 week
  Secondary evaluation index
Changes in total dosage of sublingual nitroglycerin buccal tablets | 12 weeks ± 1 week
  Secondary evaluation index
Changes of angina pectoris classification in CCS | 12 weeks ± 1 week
  Secondary evaluation index
Incidence of major cardiovascular events (MACE) | 12 weeks ± 1 week
  Secondary evaluation index
the incremental cost-effectiveness ratio (ICER) was used as the evaluation index | 12 weeks ± 1 week
  Pharmacoeconomic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Chun Liang, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He Z, Li N, Zhang W, Meng X, Wang J, Gong L, Liu B, Zheng M, Shang Z, Xu J, Jiang P, Zhao Q, Xu B, Liang C. Efficacy and safety of Shexiang Baoxin Pill in patients with angina and non-obstructive coronary arteries: A multicenter, randomized, double-blind, placebo-controlled, phase Ⅳ clinical trial. Phytomedicine. 2025 Apr;139:156556. doi: 10.1016/j.phymed.2025.156556. Epub 2025 Feb 23. PMID 40020628